CLINICAL TRIAL: NCT01779232
Title: Treatment With Danazol Before Controlled Ovarian Hyperstimulation in Women With Endometriosis Undergoing IVF
Brief Title: Danazol Treatment in Endometriosis Women Before IVF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Endocrinology and Reproductive Medicine, Italy (Network)
Responsible Party: Principal Investigator, Fabio Scarpellini, Investigator, Centre for Endocrinology and Reproductive Medicine, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-09-2013
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Endometriosis; Ovarian Cysts; Infertility
Keywords: endometriosis; ivf; ovarian reserve; danazol
MeSH Terms: conditions — Endometriosis; Ovarian Cysts; Infertility; Long Qt Syndrome 3 | interventions — Danazol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Placebo Comparator): patients treated with placebo for at least 4 months before IVF attempt
  Interventions: Drug: placebo
- danazol (Active Comparator): patients treated with danazol (100mg/day)for at least 4 months before IVF attempt
  Interventions: Drug: Danazol

INTERVENTIONS:
Drug: Danazol — 100 mg day for 4 monthh in women with diagnosed endometriosis before IVF
  Other Names: Danatrol
  Arms: danazol
Drug: placebo — administered daily like the active comparator
  Arms: control

SUMMARY:
The purpose of this study is to determine whether pre-treatment with danazol for at least 4 months before controlled ovarian hyperstimulation for IVF cycles improves pregnancy rate.

DETAILED DESCRIPTION:
Endometriosis is a chronic benign disease defined by the presence of endometrial tissue outside the uterine cavity, affecting women in their reproductive age. This disease is clinically characterized by infertility pelvic pain and the presence of ovarian cysts, endometriomas, and affects the about 10% of women. Women with endometriosis when undergo IVF show lower pregnancy rate than general population, and a reduced ovarian reserve, due to the diseases and often to ovarian surgery. The aim of this study is to evaluate if a pre-treatment with danazol, an anti-estrogenic agent, may improve the otcome of IVF cycles in these women

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of endometriosis previous laparoscopic surgery for ovarian endometriotic cysts infertility

Exclusion Criteria:

- age more than 40 years systemic disease antimulleran hormone (AMH)<1 and FSH>20

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2012-10; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 12 months
  number of ongoing pregnancy for the number of IVF cycles

SECONDARY OUTCOMES:
implantation rate | 12 months
  number of embryos implanted for the total number of embryos transferred

OTHER OUTCOMES:
number of mature oocyte collected | 12 months
  number of mature oocyte collected for patient undergoing IVF

CONTACTS AND LOCATIONS:
Overall Officials: Marco Sbracia, MD, Study Chair — Centre for Endocrinology and Reproductive Medicine, Italy
Locations (1):
- CERM, Rome, Italy